CLINICAL TRIAL: NCT02634905
Title: A Multicenter Randomized Control Trial in Children With Moderate to Severe Atopic Dermatitis to Assess the Benefit of a Nurse-led One-to-one Education Program in Addition to Standard Care Compared to Standard Care Alone on the Long Term Control of Disease Severity at 6 Months
Acronym: EDUDA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of recruitment
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC15_0035
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2021-04

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; Therapeutic patient education; pediatric dermatology
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual session therapeutic education (Experimental): The children included in the active arm will undergo, along with their parents (by child's age and wish), a structured individual TPE session between W0 and W2. This session will be conducted by the nurse trained in TPE. The session will be one hour long.
  Interventions: Other: Individual session therapeutic education; Other: Phone Call
- Control (No Intervention)

INTERVENTIONS:
Other: Individual session therapeutic education — within 2 weeks after inclusion (week 0)
  Arms: Individual session therapeutic education
Other: Phone Call
  Other Names: within 2 weeks after session therapeutic education
  Arms: Individual session therapeutic education

SUMMARY:
* Atopic dermatitis is a chronic relapsing disease, which is highly prevalent in children (15%). Therapeutic patient education (TPE) has been recognized as a key priority topic for future AD research. The strongest evidence in favour of TPE efficacy in AD comes from a large study assessing repeated multi-disciplinary group education sessions in a hospital setting. However, this type of intervention is both resource and time consuming and is not adapted to typical French practice. However, in some french dermatology centers, simple "first level" nurse-led TPE interventions are offered in addition to physicians consultations. Unfortunately, the content of these interventions seems to vary greatly depending on the caregiver and the center and the benefits of these practices have not yet been assessed. Therefore, nurse-led TPE is not considered as current care in France for AD patients.
* Thus, there is a need to rigorously assess the benefits of additional, well-structured, simple nurse-led individual TPE interventions for children with AD and their families compared to standard care alone. This study will be the first large, adequately powered, multicenter RCT trial assessing this type of intervention in children with AD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with AD, defined according to the criteria of the United Kingdom Working Party : AD should be diagnosed when a child has an itchy skin condition plus three or more of the following: Protocol EDU DA RC15_0035 Version n°4 du 15/09/16 Page 28 sur 44 CONFIDENTIAL Visible flexural dermatitis involving the skin creases, such as the bends of the elbows or behind the knees (or visible dermatitis on the cheeks and/or extensor areas in children aged under 10 years) Personal history of flexural dermatitis (or dermatitis on the cheeks and/or extensor areas in children under 10 years) Personal history of dry skin in the last 12 months Personal history of asthma or allergic rhinitis (or history of atopic disease in a firstdegree relative of children aged under 4 years)
* Onset of signs and symptoms under the age of 2 years (this criterion should not be used in children aged less than 4 years). Patient aged at least 3 months and less than 18 years.
* SCORAD 20 (moderate to severe AD)
* Patient who received treatment an anti-inflammatory topical treatment (topical corticosteroid or topical tacrolimus)
* Informed consent of parents
* Agreement of the child when appropriate
* Patient affiliated to French social security system

Exclusion Criteria:

* Patient does not meet the criteria of AD
* SCORAD < 20
* Patient aged 18 years or more
* Patient treated with oral corticosteroids currently or systemic immunosuppressant 2 months prior to the eligibility assessment
* Patients with primary immunodeficiency diseases.
* Consent not given
* Patient not affiliated to French social security system
* Patient with intercurrent disease, may be excluded if the investigator believes participation in the trial is not in the best interest of the patient
* Personal decision of the child or their parents not to be included
* Child and / or parents lack the mental capacity to give informed consent
* Child / Parents do not have a sufficient command of the French language for understanding TPE program.
* Patient or parent who has already received structured TPE for AD.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 178 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
difference in the area under the curve of SCORAD | Week 0, week 4, week 12 and week 24

SECONDARY OUTCOMES:
difference in the self-assessed long term control of disease severity measured by the area under the curve of the performed PO-SCORAD | weekly during 24 weeks
  To assess the impact of a nurses-led TPE program on Self-assessed long term control of AD severity measured using a self-assessment severity score (PO-SCORAD : patient-oriented SCORAD)
difference in disease severity measured, throughout the study by EASI | Week 0, week 4, week 12 and week 24
  To assess the impact of a nurses-led TPE program on AD severity measured by the Eczema Area and Severity Index (EASI)
difference in quality of life of the child, measured throughout the study using an age appropriate score | Week 0, week 4, week 12 and week 24
  To assess the impact of a nurses-led TPE program on Children and family quality of life.
  (Age appropriate score = IDLQI for children under 4 years old, CDLQI for children and adolescents between 4 and 18 years old)
difference in adherence to treatment measured throughout the study with the VAS scale | Week 0, week 4, week 12 and week 24
  To assess the impact of a nurses-led TPE program on Adherence to topical anti-inflammatory treatments
difference in patients/parents satisfaction assessed by a Likert scale | at week 24
  To assess the impact of a nurses-led TPE program on Parents/patients satisfaction
difference in corticosteroid phobia measured by TOPICOP score | Week 0, week 4, week 12 and week 24
  To assess the impact of a nurses-led TPE program on corticophobia

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien BARBAROT, Dr, Study Director — Nantes University Hospital
Locations (11):
- France (11):
  - Chu Bordeaux, Bordeaux
  - Chru Brest, Brest
  - Groupe Hospitalier de L Institut Catholique de Lille, Lille
  - Hospices Civils, Lyon
  - AP-HM, Marseille
  - Chu Montpellier, Montpellier
  - Chru Nancy, Nancy
  - Chu Nantes, Nantes
  - CHU NICE, Nice
  - Chu Rennes, Rennes
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No